CLINICAL TRIAL: NCT01125137
Title: Case-control Study on Matrix Metalloproteinase Levels in Tissue in Patients With Keloid Scar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Iltefat Hamzavi, Dermatologist, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB #5890
Record Dates: First submitted 2010-02-02; First posted 2010-05-18 (Estimated); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Keloid
Keywords: Keloid; MMP; Matrix metalloproteinase; dermatology
MeSH Terms: conditions — Keloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Biopsy (Experimental)
  Interventions: Procedure: Removal of Keloid

INTERVENTIONS:
Procedure: Removal of Keloid — Keloid will be excised by Henry Ford Hospital Dermatologist, Dermatosurgeon or Plastic Surgeon.

SUMMARY:
Purpose:

To compare the levels of matrix metalloproteinase-1 (MMP-1), MMP-8, MMP-13 and tissue inhibitor of metalloproteinases (TIMPs) in keloid skin tissue with normal skin in the same patient and with normal discarded skin tissue (control). The investigators aim to correlate between levels of MMPs in patients with keloid scarring in comparison with normal and discarded tissue.

DETAILED DESCRIPTION:
The investigators anticipate enrolling 20 patients into our study. The COST of the excision and related procedures WILL NOT be covered by the research study. Patient and patient's health insurance provider will be responsible for all costs of treatment and related procedures.

1. Patients must be at least 18 years old and have a keloid which they will agree to have biopsied.
2. During a screening visit we will obtain determine if patient fulfills inclusion/exclusion criteria, obtain informed visit and HIPAA authorization. Demographic information and pertinent medical history will be obtained and risk factors will be explained to the patient.
3. A focused dermatological exam will be performed assessing the severity and location of the keloid as well as skin phototype of the patient.
4. A Henry Ford Hospital Dermatosurgeon will excise a biopsy of the keloid tissue and normal tissue from enrolled patients and the specimens will be sent to the lab for workup. Discarded skin samples will also be collected from Henry Ford Plastic Surgery and Dermatology department and analyzed as an additional control for normal skin. The discarded skin samples (controls) will be region specific and matched with a keloid sample that is from the same area of the body as the biopsy sample.
5. Levels of MMP's will be measured in keloid, normal tissue samples and discarded skin samples.
6. Levels of TIMPs will be measured in keloid, normal tissue and discarded tissue samples

ELIGIBILITY:
Inclusion Criteria:

* For inclusion, the subject must:

  1. Be at least 18 years old;
  2. Have a keloid and accept to have it excised;
  3. Be able to understand the requirements for the study, the risks involved and are able to sign the informed consent form;
  4. Agree to follow and undergo all study-related procedures

Exclusion Criteria:

* Subjects will be excluded if any of the following apply:

  1. Women who are lactating, pregnant, or planning to become pregnant;
  2. Patients with a recent history of serious systemic disease;
  3. Patients who are receiving treatment for the keloid or have received treatment in the past 1 year.
  4. Any reason the investigator feels the patient should not participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Correlate the level of matrix metalloproteinases in keloid tissue versus normal skin | One time office visit for keloid excision, there will be no follow up visits for patient. Keloid tissue will be analyzed in Henry Ford Hospital laboratory after excision.

CONTACTS AND LOCATIONS:
Overall Officials: Iltefat Hamzavi, M.D., Principal Investigator — Henry Ford Hospital
Locations (1):
- Henry Ford Hospital Dermatology Dept. 3031 West Grand Blvd, Suite 800, Detroit, Michigan, United States